CLINICAL TRIAL: NCT00173927
Title: The Differences in Images of Vertebral Artery Stenosis and Carotid Artery Stenosis Pre- and Post-Percutaneous Transluminal Angioplasty and the Gene Expression Patterns in Peripheral White Blood Cells
Brief Title: Images in Extracranial Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701156; NTUH 94N04
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2005-09

CONDITIONS: Extracranial Atherosclerosis
Keywords: extracranial atherosclerosis; imaging; biomarkers

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The goals of this trial are:

1. To compare the sensitivity and specificity of various tools including Doppler and magnetic resonance imaging (MRI) for diagnosing vertebral artery stenosis and carotid artery stenosis. The positron emission tomography (PET)/MRI fusion imaging will be a promising tool to provide both anatomical and functional imaging for vulnerable plaques.
2. To identify patients at high risk of plaque rupture by image studies, biomedical profile, and gene expression of circulating monocytes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic extracranial atherosclerosis who are going to receive angiography and possible intervention.

Exclusion Criteria:

* Acute systemic illness
* Creatinine > 3 mg/dl
* Unable to tolerate the tests (including MRI and PET/computed tomography [CT] scans)

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Li Kao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan